CLINICAL TRIAL: NCT02454387
Title: A Double-blind, Single and Multiple Ascending Dose, Randomised, Placebo-controlled Study, in Healthy Adult and Elderly Subjects Exploring Safety, Tolerability, Pharmacokinetics of ONO-4474 and Pharmacology of ONO-4474 in NGF-hyperalgesia
Brief Title: A Study to Evaluate Safety, Tolerability, Pharmacokinetics and Pharmacology of ONO-4474 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ONO-4474-01
Record Dates: First submitted 2015-04-29; First posted 2015-05-27 (Estimated); Last update posted 2016-06-30 (Estimated); Status verified 2016-01

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (10):
- Experimental: ONO-4474 Part A1 (Experimental): Single doses of ONO-4474 or placebo, randomized 3 active: 1 placebo
  Interventions: Drug: ONO-4474 Part A1
- Experimental: ONO-4474 Placebo Part A1 (Placebo Comparator): Single doses of ONO-4474 or placebo, randomized 3 active: 1 placebo
  Interventions: Drug: Placebo Part A1
- Experimental: ONO-4474 Part A2 (Experimental): Single doses (2 periods) of ONO-4474 or placebo, randomized 3 active: 1 placebo
  Interventions: Drug: ONO-4474 Part A2
- Experimental: ONO-4474 Placebo Part A2 (Placebo Comparator): Single doses (2 periods) of ONO-4474 or placebo, randomized 3 active: 1 placebo
  Interventions: Drug: Placebo Part A2
- Experimental: ONO-4474 Part B (Experimental): Multiple ascending doses of ONO-4474 or placebo, randomized 3 active: 1 placebo
  Interventions: Drug: ONO-4474 Part B
- Experimental: ONO-4474 Placebo Part B (Placebo Comparator): Multiple ascending doses of ONO-4474 or placebo, randomized 3 active: 1 placebo
  Interventions: Drug: Placebo Part B
- Experimental: ONO-4474 Part C (Experimental): NGF hyperalgesia and single or multiple doses of ONO-4474, randomized 1 active: 1 placebo in cross over design
  Interventions: Drug: ONO-4474 Part C
- Experimental: ONO-4474 Placebo Part C (Placebo Comparator): NGF hyperalgesia and single or multiple doses of ONO-4474, randomized 1 active: 1 placebo in cross over design
  Interventions: Drug: Placebo Part C
- Experimental: ONO-4474 Part D (Experimental): Single doses of ONO-4474 or placebo, randomized 3 active: 1 placebo
  Interventions: Drug: ONO-4474 Part D
- Experimental: ONO-4474 Placebo Part D (Placebo Comparator): Single doses of ONO-4474 or placebo, randomized 3 active: 1 placebo
  Interventions: Drug: Placebo Part D

INTERVENTIONS:
Drug: ONO-4474 Part A1 — Healthy volunteers
  Other Names: ONO-4474
  Arms: Experimental: ONO-4474 Part A1
Drug: Placebo Part A1 — Healthy volunteers
  Other Names: Placebo
  Arms: Experimental: ONO-4474 Placebo Part A1
Drug: ONO-4474 Part A2 — Healthy volunteers
  Other Names: ONO-4474
  Arms: Experimental: ONO-4474 Part A2
Drug: Placebo Part A2 — Healthy volunteers
  Other Names: Placebo
  Arms: Experimental: ONO-4474 Placebo Part A2
Drug: ONO-4474 Part B — Healthy volunteers
  Other Names: ONO-4474
  Arms: Experimental: ONO-4474 Part B
Drug: Placebo Part B — Healthy volunteers
  Other Names: Placebo
  Arms: Experimental: ONO-4474 Placebo Part B
Drug: ONO-4474 Part C — Healthy volunteers
  Other Names: ONO-4474
  Arms: Experimental: ONO-4474 Part C
Drug: Placebo Part C — Healthy volunteers
  Other Names: Placebo
  Arms: Experimental: ONO-4474 Placebo Part C
Drug: ONO-4474 Part D — Healthy volunteers
  Other Names: ONO-4474
  Arms: Experimental: ONO-4474 Part D
Drug: Placebo Part D — Healthy volunteers
  Other Names: Placebo
  Arms: Experimental: ONO-4474 Placebo Part D

SUMMARY:
A Phase 1 Study to Evaluate Safety, Tolerability, Pharmacokinetics and Pharmacology of ONO-4474 in healthy volunteers.

DETAILED DESCRIPTION:
A Double-blind, Multi-centre, Single Dose, Single and Multiple Ascending Dose, Four-part, Randomised, Placebo-controlled Study in Healthy Adult and Elderly Subjects Exploring the Safety, Tolerability, Pharmacokinetics of ONO-4474 in Fed and Fasted Conditions, and Pharmacology of ONO-4474 in NGF-hyperalgesia.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subjects aged 18-55 years inclusive (Parts A and C); healthy male and female subjects aged 18-55 years inclusive (Part B); healthy male and female subjects aged 65 and over (Part D)
2. Subjects with a body mass index of 18.0-30.0 kg/m2 inclusive

Exclusion Criteria:

1. Subjects who have a clinically relevant history or presence of any clinically significant disease or disorder
2. Current smokers or those that have smoked or used nicotine products within 6 months of the Screening visit

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2015-05; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of ONO-4474 across ascending single and multiple doses using number of adverse events | Up to Day 28

SECONDARY OUTCOMES:
Maximum plasma concentration of ONO-4474 (Cmax) | Day 1 and at Day 7
ONO-4474 Plasma Area Under the Curve from Time Zero to 24 hour after dosing (AUC24) | Day 1 and at Day 7
Time to Reach Maximum Observed Plasma concentration (Tmax) of ONO-4474 | Day 1 and at Day 7
Plasma Decay half life (T1/2) of ONO-4474 | Day 1 and at Day 7
Part C only - Evaluation of ONO-4474 vs. placebo on walking soreness using a Likert scale | 3hr and 24hr after NGF injection
Part C only: Assessment of pharmacology of ONO-4474 using change in pressure pain threshold after NGF injection. | 3hr and 24hr after NGF injection
  Pressure algometry at site of NGF injection (anterior tibialis)

CONTACTS AND LOCATIONS:
Overall Officials: Drug Development Division, Study Director — Ono Pharmaceutical Co. Ltd
Locations (2):
- Aalborg Clinical Site, Aalborg, Denmark
- Nottingham Clinical SIte, Nottingham, United Kingdom